CLINICAL TRIAL: NCT06625944
Title: Prospective Cohort Study to Understand Impact of Viral Infection in Chronic Lung Disease
Brief Title: Exploring How Viral Infections Affect People With Chronic Lung Disease
Acronym: PRIVILEGE
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 172663; 336487 (Other: IRAS)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Bronchiectasis Adult; Bronchiectasis With Acute Exacerbation; COPD (Chronic Obstructive Pulmonary Disease); Respiratory Infection Virus
Keywords: Natural Cohort; Prospective; Bronchiectasis; Chronic Lung Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Nasal Samples, Sputum, Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many people with chronic lung disease have disease flare-ups. It was previously believed that these were mainly caused by bacteria but recent evidence suggests that viruses could be an important trigger. This study will recruit volunteers with chronic lung disease and take samples both when well (at baseline) and during flare-ups (exacerbations) to better understand the role of viruses in triggering exacerbations and also how the immune response is affected. The researchers will follow the volunteers' progress for up to two years. Whenever they get unwell they will take some samples (nose swabs, finger prick testing, phlegm sample) and post them to the researchers. Then, they will come in for a visit for more samples (blood tests, further swabs) and a review.

DETAILED DESCRIPTION:
Individuals with chronic lung disease are characterised by exacerbations (episodes of increased symptoms such as breathlessness, sputum production etc) which have been shown to be important drivers of disease severity. Viral infections are well recognised causes of asthma exacerbations but the same detail of understanding regarding the effect of viral infection on other chronic respiratory conditions such as chronic obstructive pulmonary disease (COPD) and bronchiectasis is lacking. During the COVID-19 pandemic, when isolation measures were in place for individuals with chronic respiratory disease, episodes of exacerbation were substantially decreased, suggesting a causal link between viruses and exacerbations. Such information is critical in an age with increasing concerns regarding antibiotic resistance and may change practice towards early administration of antiviral agents for respiratory disease exacerbations. To date, prospective surveillance studies in chronic lung disease have been predominantly cross sectional and focussed on hospitalised individuals where presentation is often late with reduced sensitivity for viral detection and no understanding of baseline disease state. The our study will establish closely monitored prospective patient cohort in order to assess their viral and immune status at baseline and in the early phases of an exacerbation in order to better understand the role of respiratory viruses in chronic lung disease.

Specifically, this unique study design will allow us to study the following important areas in unprecedented detail and depth: (i) Early identification and diagnosis of clinical deterioration / exacerbations to comprehensively understand the role played by viruses in chronic lung disease exacerbations. (ii) Full capture of all clinical deterioration / exacerbation events experienced by patients with chronic lung disease including mild, typically unreported episodes. (iii) Evaluation of the immune and microbiological dynamics associated with recovery from exacerbation episodes and the impact upon longer term disease progression.

Clinical Visits and Sampling:

(i) Baseline study visit: All eligible individuals will undergo screening when clinically stable including clinical history/ examination, respiratory function testing (spirometry) and a severity assessment with the use of validated questionnaires (COPD assessment test (CAT), Bronchiectasis Health Questionnaire (BHQ)). Clinical information including microbiology cultures, the underlying lung disease and other medical conditions and medication history will be obtained from medical records.

Prior imaging including CT images will be pseudoanonymised and stored for radiological scoring and analysis. At the first study visit the following biological samples will be taken to address the study objectives:

* sputum
* nasal samples (Nasopharyngeal swab, synthetic absorptive matrix (SAM) sampling to sample nasal lining fluid and nasal brushings)
* Exhaled breath
* Venous (40mls) and capillary blood (~0.5mls)
* Stool (remote stool sampling (performed at home and posted in) using secure bespoke collection kits)

(ii) Exacerbation monitoring and sampling: All participants will record daily diary cards which will be monitored by the study team. This will enable full characterisation of all exacerbations including those that would typically be unreported in routine clinical circumstances. Participants that develop symptoms of acute viral infection or acute exacerbation will have the following sampling and clinical assessment as detailed above.

* Early exacerbation sampling (<48hrs of increased symptoms) (REMOTE STUDY VISIT from home)
* Remote nasopharyngeal swab and sputum sampling with bespoke collection kits
* Remote capillary blood sampling with bespoke collection kits
* Mid-exacerbation sampling (within 5 days of increased symptoms) (IN PERSON VISIT)
* clinical assessment, spirometry, validated questionnaires (as per baseline)
* sputum
* nasal samples (Nasopharyngeal swab, SAM and nasal brushings)
* Exhaled breath
* Venous (40mls) and capillary blood (~0.5mls)
* Stool (remote stool sampling using bespoke collection kits)
* Exacerbation recovery sampling (4 weeks after initial increased symptoms) (REMOTE STUDY VISIT from home)
* Remote nasopharyngeal swab, SAM and sputum sampling with bespoke collection kits
* Remote capillary blood sampling with bespoke collection kits (iii) Stable longitudinal assessment: All participants will undergo further clinical visits similar to baseline at 12 monthly intervals over a 2 year period (as detailed above)

ELIGIBILITY:
Inclusion Criteria:

* Adults with a physician confirmed diagnosis of chronic airway disease (e.g. COPD and bronchiectasis) according to established diagnostic criteria.

AND

- Prior history of exacerbation within last year (defined as requiring antibiotic and/or corticosteroids).

Exclusion Criteria:

* Inability to complete daily symptom diaries and/or attend for clinical assessments.
* Exacerbation within 4 weeks of study recruitment and/or clinical instability at the time of recruitment.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lung disease under the care of respiratory teams at Royal Brompton and Harefield (NHS) Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Respiratory viruses detection during exaccerbations | All exacerbations within a 24 month follow up period.
  The percentage of chronic airway disease exacerbations where a respiratory virus is detected (with sub-classification of the specific viral subtypes).

SECONDARY OUTCOMES:
Differences in symptoms between viral and non-viral exacerbations | All exacerbations within a 24 month follow up period.
  Differences in magnitude of deterioration in symptoms (as measured by validated symptom score) between viral and non-viral exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Shah, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No